CLINICAL TRIAL: NCT04439643
Title: Plaque Stratification Using Ccta in Coronary ARtery Disease (PoSTCARD)
Acronym: PoSTCARD
Status: Completed | Type: Observational
Sponsor: Elucid Bioimaging Inc. (Industry)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: PoSTCARD
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Development / training: Selected by stratified partitioning
  Interventions: Device: vascuCAP
- Sequestered / test: Selected by stratified partitioning
  Interventions: Device: vascuCAP

INTERVENTIONS:
Device: vascuCAP — time to event and phenotype classification model

SUMMARY:
Develop time-to-event prediction and plaque phenotype classification models for patients with known or suspected coronary artery disease.

DETAILED DESCRIPTION:
Develop time-to-event prediction and plaque phenotype classification models using plaque morphology and composition assessment of CTA which has been validated by histology, applied to representative cohort of patients. Generalizability of models is enhanced by using validated rather than only raw image inputs. Demographic, clinical, and outcome data is collected for enrolled patients as well as last known well dates.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have successfully completed at least one (possibly multiple) CCTA for known or suspected coronary artery disease, which was positive for coronary atherosclerotic changes.
* Subject must have been ≥ 18 years of age at the time of the CCTA

Exclusion Criteria:

* Subject has a history of percutaneous coronary intervention (PCI) with stent implantation and/or coronary artery bypass grafting (CABG)
* CCTA taken less than 3 months after deployment of new scanner
* Subject with insufficient CCTA image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Reverse chronological, all-comers, design, adjusted for demographic factors
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Time to adverse outcome | >= 2 years
  Develop time-to-event model for major adverse cardiac events (MACE) prediction on large retrospective cohort (and enable a prospective collection subsequent to this study). Consistent with this primary endpoint is the evaluation of all imaging-derived data that has a bearing on the diagnosis and prognosis of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Buckler, MS, Principal Investigator — Elucid Bioimaging Inc.
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No